CLINICAL TRIAL: NCT07073157
Title: Effect of HRS-8427 for Injection on the Pharmacokinetics of Furosemide and Metformin in Healthy Subjects。
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HRS-8427-106
Record Dates: First submitted 2025-06-30; First posted 2025-07-18 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-06

CONDITIONS: Health Volunteer
MeSH Terms: interventions — Furosemide; Metformin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HRS-8427 injection plus furosemide (Experimental)
  Interventions: Drug: HRS-8427 injection plus furosemide
- HRS-8427 injection plus metformin (Experimental)
  Interventions: Drug: HRS-8427 injection plus metformin

INTERVENTIONS:
Drug: HRS-8427 injection plus furosemide — HRS-8427 injection plus furosemide
  Arms: HRS-8427 injection plus furosemide
Drug: HRS-8427 injection plus metformin — HRS-8427 injection plus metformin
  Arms: HRS-8427 injection plus metformin

SUMMARY:
The pharmacokinetics of HRS-8427 for injection on the transporter OAT1 substrate furosemide and the MATE1/METE2-K substrate metformin were evaluated in healthy subjects. The safety of HRS-8427 for injection was evaluated in combination with furosemide and metformin.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male and female subjects aged from 18 to 45 years old (including 18 and 45 years old, subject to the time of signing the informed consent)
2. Body weight ≥45 kg for female subjects and ≥50 kg for male subjects with body mass index (BMI) in the range of 19.0-26.0 kg/m2 (BMI = weight (kg)/height 2 (m2)), including boundary values
3. Female subjects were not pregnant or lactating and had a negative pretrial pregnancy test. Male or female subjects agreed to use a highly effective contraceptive method approved by the investigator as required by the investigator (see Appendix 13 to the protocol) for the duration of the trial, with no sperm/egg donation planned (from the time of informed consent until 3 months after the last dose).
4. have understood the nature, significance, possible benefits, possible inconvenience and potential risks of the trial in detail before the trial, and voluntarily participate in the clinical trial, can communicate well with the investigators, comply with the requirements of the whole study, and sign the written informed consent

Exclusion Criteria:

1. Have a history of food or drug allergy
2. previous or current diseases of the heart, liver, kidney, endocrine, digestive tract, immune system, respiratory system, musculoskeletal system, and nervous system
3. Plasma concentrations of sodium, potassium, magnesium and calcium were lower than the normal range and serum creatinine was not in the normal range
4. Patients with fasting blood glucose below the normal range or a history of hypoglycemia.
5. Abnormal 12-lead electrocardiogram and the investigator's judgment that the patient is not suitable for the study (including but not limited to QTcF > 450 ms, severe arrhythmia such as atrioventricular block of degree II or above)
6. Laboratory tests (blood routine test, urine routine test, urine sediment test, blood biochemistry, coagulation function test, thyroid function test), physical examination, vital signs (temperature, blood pressure, pulse), abdominal ultrasound and chest X-ray results were judged by clinicians as clinically significant abnormalities。
7. Infectious disease tests (human immunodeficiency virus antibody, hepatitis B surface antigen, anti-hepatitis C virus antibody, anti-treponema pallidum specific antibody) were positive。
8. Patients who underwent major surgery within 3 months before screening; Or underwent surgery that may affect the in vivo course or safety evaluation of the study drug; Or planned to undergo surgery during the study period。
9. Participants who had been enrolled in a drug clinical trial within 3 months before screening and had taken a trial drug, or who planned to participate in another clinical trial during the study period。
10. Participants who had donated blood or had a blood loss of more than 300 mL or received a transfusion or blood product within 3 months before screening or were scheduled to donate blood during or within 1 month after the trial。
11. Those who had a history of drug abuse within 3 months before screening, had a history of drug use, or had a positive screening test for drug abuse。
12. The participant had any other factor that was deemed by the investigator to preclude participation in the trial

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2025-07-15 (Actual); Primary Completion 2025-08-15 (Actual); Study Completion 2025-08-15 (Actual)

PRIMARY OUTCOMES:
Cmax | The observation lasted until the 9th day
AUC0-t | The observation lasted until the 9th day
AUC0-∞ | The observation lasted until the 9th day
Tmax | The observation lasted until the 9th day
t1/2 | The observation lasted until the 9th day
CL/F | The observation lasted until the 9th day
Vz/F | The observation lasted until the 9th day

SECONDARY OUTCOMES:
adverse events | The observation lasted until the 16th day

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Fujian Medical University, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: Undecided